CLINICAL TRIAL: NCT00985816
Title: The Effects of Lactobacillus Reuteri DSM 17938 on Immunomodulation and Gastric Motility in Preterm Newborns
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: University of Bari Departement of Pediatrics, Flavia Indrio
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FI-LR2009
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2009-09

CONDITIONS: Preterm Birth
Keywords: Preterm; newborns; Gastric; Motility; Mucosal; immunity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L reuteri DSM 17938 (Active Comparator): L. reuteri DSM 17938 will be given at a dose of 1x108 colony forming units (CFU)/day in an oil formulation delivered from a drop bottle. In the active study product, freeze-dried L. reuteri is suspended in a mixture of pharmaceutical grade medium chain triglycerides and sunflower oil together with pharmaceutical grade silicon dioxide to give the product the correct rheological properties (Connolly, 2005). The placebo consists of an identical formulation except that the L. reuteri is not present. This dose of the oil formulation with L. reuteri has been shown to induce significant colonisation in infants and is well-tolerated (Abrahamsson et al., 2007; Savino et al., 2007; Indrio et al., 2008).
  Interventions: Dietary Supplement: Lactobacillus Reuteri
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus Reuteri — L. reuteri DSM 17938 will be given at a dose of 1x108 colony forming units (CFU)/day
  Arms: L reuteri DSM 17938
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The investigators propose a Phase II interventional trial to investigate the role of Lactobacillus reuteri DSM 17938 on the intestinal motility and immune response of premature infants and further evaluate safety of the use of this probiotic in a population of premature infants.

DETAILED DESCRIPTION:
Hypothesis Administration of Lactobacillus reuteri to premature infants will improve their intestinal motility when compared with infants receiving placebo. Primary Objective Evaluate the effects of L. reuteri in the intestinal motility by measuring the gastric emptying rate in infants before and after 21 consecutive days of administration of L. reuteri.

Secondary Objectives 1. Mechanisms of action of L. reuteri - L.reuteri impact in the host immune response by determining fecal cytokines, sIgA and calprotectin before and after 21 days of administration - L.reuteri rate of colonization after its administration.

2. Efficacy and safety of L. reuteri to premature infants - Clinical beneficial effects secondary to the administration of L. reuteri to premature infants. The following clinical outcomes will be identified and compared between groups:

* Number of gastrointestinal symptoms (regurgitation, vomiting, stasis)
* Days to full feeds. Number of days to reach full feeds defined as > 120cc/kg/day) x2 days or more.
* Days on parenteral nutrition
* Weight gain defined as the number of days needed to reach 150% of birth weight
* Length of hospital stay
* Any possible side effects and adverse events secondary to the administration of L. reuteri to premature infants.
* Incidence of late onset sepsis.
* Incidence and severity of necrotizing enterocolitis categorized by Bell's classification
* Use of antibiotics (number of days on antibiotics during the hospital stay)
* Mortality (at 28 days after birth and at hospital discharge).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 30 - 32 weeks. Gestational age will be defined by the best estimate based on prenatal ultrasound in the first trimester, DLM and/or Balard Score after birth.

Exclusion Criteria:

* Cardiovascular or (respiratory) instability after 48 hours of age - Chromosomal anomalies.
* Major congenital anomalies (complex cardiac anomalies, congenital hydrocephalus, renal dysplasia)
* Congenital (e.g. jejunal atresia) and acquired (e.g. GI perforation) gastrointestinal pathology precluding oral feed and/or requiring major surgical or medical intervention
* Parental refusal
* Prior enrollment into a conflicting clinical trial. Conflicting clinical trial will be those in which the intervention could modify the outcome of the present study, for example studies that could alter the intestinal motility or the immune response of the premature infants.

Ages: 3 Days to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of L. reuteri in the intestinal motility by measuring the gastric emptying rate in infants before and after 21 consecutive days of administration of L. reuteri | 21 days

SECONDARY OUTCOMES:
Mechanisms of action of L.reuteri | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Indrio, Principal Investigator — University of Bari
Locations (1):
- Flavia Indrio, Bari, Italy